CLINICAL TRIAL: NCT00381095
Title: A Randomized Placebo-Controlled Trial Of The Efficacy And Tolerability Of Flexibly Dosed Pregabalin In The Treatment Of Cancer-Induced Bone Pain
Brief Title: A Study To Evaluate Pregabalin In The Treatment Of Moderate To Severe Chronic Bone Pain Related To Metastatic Cancer
Acronym: COPE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0081128
Record Dates: First submitted 2006-09-25; First posted 2006-09-27 (Estimated); Results first posted 2011-09-27 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2019-04

CONDITIONS: Bone Neoplasms; Pain, Intractable; Cancer
MeSH Terms: conditions — Bone Neoplasms; Pain, Intractable; Neoplasms | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): flexible dosing
  Interventions: Drug: Pregabalin
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin — Capsule, Flexible-dosing, Double-blind. Treatment duration is 28 days at 100-600 mg/day administered BID+ taper (6 days).
  Arms: 1
Drug: Placebo — Placebo
  Arms: 2

SUMMARY:
The purpose of this study is to assess the analgesic efficacy of flexibly-dosed pregabalin in the adjunctive treatment of subjects with cancer-induced bone pain.

DETAILED DESCRIPTION:
Pfizer decided to discontinue additional enrollment into the study effective Sept 5 2010 after assessing the feasibility of completing this study in a realistic timeframe.The study was not stopped for any safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a malignant, solid tumor that has been diagnosed as having metastasized to bone, and must have moderate to severe pain secondary to the bone metastasis at an identifiable reference site.

Exclusion Criteria:

* The patient who has undergone diagnostic or therapeutic invasive interventions (angiography, biopsy, surgery) less than 15 days prior to study start that would impact their assessment of pain at the reference pain site or area, in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2006-12; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (50):
- United States (7):
  - Pfizer Investigational Site, Celebration, Florida
  - Pfizer Investigational Site, Kissimmee, Florida
  - Pfizer Investigational Site, Pensacola, Florida
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Edina, Minnesota
  - Pfizer Investigational Site, Canton, Ohio
  - Pfizer Investigational Site, Dover, Ohio
- Pfizer Investigational Site, Hamilton, Ontario, Canada
- Czechia (6):
  - Pfizer Investigational Site, Benesov U Prahy
  - Pfizer Investigational Site, Hořovice
  - Pfizer Investigational Site, Jablonec nad Nisou
  - Pfizer Investigational Site, Pilsen
  - Pfizer Investigational Site, Praha 1 - Nove Mesto
  - Pfizer Investigational Site, Praha 6 - Hradcany
- Pfizer Investigational Site, Cairo, Egypt
- Finland (2):
  - Pfizer Investigational Site, Helsinki
  - Pfizer Investigational Site, Joensuu
- France (2):
  - Pfizer Investigational Site, Bordeaux
  - Pfizer Investigational Site, Villejuif
- Hungary (4):
  - Pfizer Investigational Site, Budapest
  - Pfizer Investigational Site, Nyíregyháza
  - Pfizer Investigational Site, Szentes
  - Pfizer Investigational Site, Tata
- Italy (2):
  - Pfizer Investigational Site, Aviano (PN)
  - Pfizer Investigational Site, Milan
- Mexico (2):
  - Pfizer Investigational Site, Monterrey, Nuevo León
  - Pfizer Investigational Site, México D.F
- Pfizer Investigational Site, Lima, Peru
- Philippines (2):
  - Pfizer Investigational Site, Manila
  - Pfizer Investigational Site, Quezon City
- Poland (5):
  - Pfizer Investigational Site, Bialystok
  - Pfizer Investigational Site, Gdansk
  - Pfizer Investigational Site, Kielce
  - Pfizer Investigational Site, Lodz
  - Pfizer Investigational Site, Warsaw
- Russia (3):
  - Pfizer Investigational Site, Vsevolozhsk, Vsevolozhsk District, Leningrad Region
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Saint Petersburg
- South Korea (2):
  - Pfizer Investigational Site, Daegu
  - Pfizer Investigational Site, Seoul
- Spain (2):
  - Pfizer Investigational Site, Alcorcón, Madrid
  - Pfizer Investigational Site, Lleida
- Sweden (2):
  - Pfizer Investigational Site, Örebro
  - Pfizer Investigational Site, Stockholm
- Taiwan (3):
  - Pfizer Investigational Site, Kaohsiung Hsien
  - Pfizer Investigational Site, Taichung
  - Pfizer Investigational Site, Taipei
- Thailand (2):
  - Pfizer Investigational Site, Rachathewi, Bangkok
  - Pfizer Investigational Site, Ratchathewi, Bangkok
- Pfizer Investigational Site, Caracas, Distrito Federal, Venezuela

REFERENCES:
- [Derived] Sjolund KF, Yang R, Lee KH, Resnick M. Randomized study of pregabalin in patients with cancer-induced bone pain. Pain Ther. 2013 Jun;2(1):37-48. doi: 10.1007/s40122-013-0009-8. Epub 2013 Feb 26. PMID 25135035
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081128&StudyName=A%20Study%20To%20Evaluate%20Pregabalin%20In%20The%20Treatment%20Of%20Moderate%20To%20Severe%20Chronic%20Bone%20Pain%20Related%20To%20Metastatic%20Cancer

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A0081128 terminated on 01-SEP-2010 due to slow enrollment, analysis at 50 percent (%) enrollment determined that increasing the sample size would require significant extension of enrollment period.
Groups:
- Pregabalin: Pregabalin Flexible Dose 50 to 300 milligrams (mg) capsules orally twice per day (100 to 600 mg/day) for 28 days. Dose adjustments from Day 2 up to Day 14 as needed, followed by fixed dosing through Day 28, followed by dose tapering to Day 34
- Placebo: Matching placebo capsules orally twice per day
Period: Overall Study
Arm/Group | Pregabalin | Placebo
Started | 72 | 80
Completed | 59 | 59
Not Completed | 13 | 21
Not completed — Death | 3 | 4
Not completed — Lack of Efficacy | 2 | 4
Not completed — Other | 2 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Adverse Event | 2 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin | Placebo | Total
Number analyzed (Participants) | 72 | 80 | 152
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 54 | 104
  >=65 years | 22 | 26 | 48
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 41 | 77
  Male | 36 | 39 | 75

OUTCOME MEASURES:

1. Primary Outcome: Duration Adjusted Average Change (DAAC) From Baseline in Daily Worst Pain, Fixed Dosing Date to Day 28
Description: DAAC from baseline based on Numeric Rating Scale (NRS) score for Worst Pain at Reference site from the last day dose adjustment was needed (fixed dosing date) to day 28. DAAC defined as area under the curve (AUC) of change in worst pain divided by pain measurement duration. Pain rated on an 11 point scale ranged from 0 (no pain) to 10 (worst possible pain). Change was week x minus baseline.
Time Frame: Baseline, Fixed Dosing Date to Day 28 or Early Termination (ET)
Population: Intent-To-Treat population (ITT): all randomized participants for whom at least one post-baseline efficacy evaluation was obtained; N= the number of participants with evaluable data analyzed; n= number of participants with evaluable data at the specific time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 72 | 79
Units on a scale
  Baseline (n=72, 79) | 6.28 (1.68) | 6.47 (1.59)
  Change at Day 28 (n=72, 77) | -1.53 (1.81) | -1.23 (1.74)

2. Secondary Outcome: DAAC From Baseline in Daily Worst Pain, Days 1 Through 28
Description: DAAC from baseline in the daily worst pain based on the NRS Worst Pain at Reference Site score collected from participant's daily diary. Pain rated on an 11 point scale ranged from 0 (no pain) to 10 (worst possible pain). DAAC defined as AUC of daily worst pain score divided by pain measurement duration. Change was week x minus baseline.
Time Frame: Baseline, Days 1 through 28 or ET
Population: ITT; N= number of participants with evaluable data analyzed
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 72 | 77
Units on a scale | -1.27 (1.45) | -1.03 (1.37)

3. Secondary Outcome: DAAC From Baseline in Daily Worst Pain, Day 1 to End of Dose Adjustment
Description: as for outcome 2
Time Frame: Baseline, Day 1 to End of Dose Adjustment or ET
Population: ITT; N= number of participants with evaluable data analyzed
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 69 | 76
Units on a scale | -0.72 (1.11) | -0.53 (1.01)

4. Secondary Outcome: DAAC From Baseline in Daily Worst Pain 14 Days After Fixed Dosing Date Up to Day 28
Description: DAAC from baseline in the daily worst pain based on the NRS Worst Pain at Reference Site score collected from participant's daily diary 14 days after dosing stabilized (fixed dosing date) up to Day 28. Pain rated on an 11 point scale ranged from 0 (no pain) to 10 (worst possible pain). DAAC defined as AUC of daily worst pain score divided by pain measurement duration. Change was week x minus baseline.
Time Frame: Baseline, 14 Days After Fixed Dosing Date up to Day 28 or ET
Population: ITT; N= number of participants with evaluable data analyzed
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 72 | 77
Units on a scale | -1.47 (1.79) | -1.15 (1.72)

5. Secondary Outcome: Change From Baseline in Modified Brief Pain Inventory (mBPI-sf) Pain Severity Index Score at Week 4
Description: m-BPI-sf: participant rated 11-point Likert rating scale ranging from 0 (no pain) to 10 (worst pain possible). Pain severity index was the mean of item scores 1, 2, 3, and 4 (worst, least, average and current pain scores). Change was scores at observation minus scores at baseline.
Time Frame: Baseline, Week 4 or ET
Population: ITT; LOCF= Last observation carried forward; n= number of evaluable participants analyzed at each time point; N= number of participants with evaluable data analyzed
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 71 | 77
Units on a scale
  Baseline (n=71, 77) | 5.18 (1.80) | 5.03 (1.72)
  Change at Week 4 (n=59, 59) | -2.06 (1.75) | -1.41 (2.51)
  Change at Week 4/LOCF (n=64, 63) | -1.94 (1.88) | -1.35 (2.54)

6. Secondary Outcome: Change From Baseline in mBPI-sf Interference Index Score at Week 4
Description: m-BPI-sf: participant-rated 11 point Likert rating scale ranging from 0 (does not interfere) to 10 (completely intereres) with functional activities (general activity, mood, walking ability, relations with other people, sleep, normal work, and enjoyment of life) in past 24 hours. Change was score at each observation minus baseline score.
Time Frame: Baseline, Week 4 or ET
Population: ITT; LOCF; n= number of evaluable participants analyzed at each time point; N= number of participants with evaluable data analyzed
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 71 | 76
Units on a scale
  Baseline (n=71, 76) | 4.92 (2.22) | 5.27 (2.14)
  Change at Week 4 (n=59, 58) | -1.83 (2.47) | -1.50 (2.44)
  Change at Week 4/LOCF(n=64, 62) | -1.66 (2.57) | -1.48 (2.56)

7. Secondary Outcome: Change From Baseline in Average Pain Scores at Weeks 1, 2, 3 and 4
Description: Change from baseline in daily average pain score NRS 0 (no pain) to 10 (pain as bad as you can imagine) for pain intensity over past 24 hours recorded every evening before bedtime. Change was week x average minus baseline average.
Time Frame: Baseline, Weeks 1, 2, 3 and 4 or ET
Population: Data not analyzed due to early study termination.
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change From Baseline in Total Daily Dose of Opioids Day 0 Through Day 28
Description: Change from baseline in total daily dose of opioids immediate release (IR), sustained release (SR) formulations separately and combined.
Time Frame: Baseline, Day 0 through Day 28 or ET
Population: Data no analyzed due to early study termination.
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change From Pre-Baseline in Total Daily Dose of Morphine Equivalents Day 0 Through Day 28
Description: IR and SR formulations separately and combined. Change was day x minus baseline.
Time Frame: Baseline, Day 0 through Day 28 or ET
Population: Data not analyzed due to early study termination.
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression Scale (HADS) at Week 4
Description: HADS: participant rated questionnaire with 2 subscales. HADS-Anxiety assessed generalized anxiety (anxious mood/ restlessness/ anxious thoughts/panic attacks); HADS-Depression assessed lost interest/diminished pleasure response (lowering of hedonic tone). Each subscale has 7 items which ranged from 0 (no presence of anxiety or depression) to 3 (severe feeling anxiety/depression). Total 0-21 for each subscale; higher score indicates greater severity of anxiety and depression symptoms. Change was week x minus baseline.
Time Frame: Baseline, Week 4 or ET
Population: ITT; LOCF; n= number of evaluable participants analyzed at each time point; N= number of participants with evaluable data analyzed; individual symptoms not analyzed
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 72 | 78
Units on a scale
  Anxiety Baseline (n= 72, 78) | 11.61 (2.94) | 11.60 (2.74)
  Anxiety Change at Week 4 (n= 60, 60) | 0.98 (3.31) | 0.80 (2.29)
  Anxiety Change at Week 4/LOCF (n=64, 65) | 0.80 (3.37) | 0.71 (2.42)
  Depression Baseline (n= 72, 78) | 9.33 (2.18) | 10.15 (2.59)
  Depression Change at Week 4 (n= 60, 60) | 0.20 (2.77) | -0.57 (2.13)
  Depression Change at Week 4/LOCF (n=64, 65) | 0.22 (2.73) | -0.57 (2.81)

11. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: PGIC: participant rated instrument to measure participant's change in overall status on a 7-point scale; range from 1 (very much improved) to 7 (very much worse).
Time Frame: Weeks 2 and 4 or ET
Population: ITT; LOCF; n=number of evaluable participants analyzed at each time point; N= the number of participants with evaluable data analyzed
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 69 | 74
Units on a scale
  Week 2 (n=66,68) | 2.97 (1.36) | 3.09 (1.19)
  Week 4 (n=59, 60) | 2.73 (1.39) | 2.87 (1.46)
  LOCF/ET (n=69, 74) | 2.88 (1.46) | 2.99 (1.45)

12. Secondary Outcome: Change From Baseline in Opioid-Related Symptoms Distress Scale (OR-SDS) at Day 14 and Day 28
Description: OR-SDS included OR-SDS individual items by dimension of frequency (rarely to almost constantly), severity (slight to very severe), and degree of bother (not at all to very much), number of episodes of retching/vomiting, OR-SDS dimension composite and overall composite scores. Change was scores at occurance minus score at baseline.
Time Frame: Baseline, Day 14, Day 28 or ET
Population: Data not analyzed due to early study termination.
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Change From Baseline in Eastern Cooperative Oncology Group Performance (ECOG) Status Scale at Day 28
Description: ECOG - assessed disease progression and how disease affected the daily living abilities of the participant and determined appropriate treatment and prognosis. Graded 0 (fully active able to carry on all pre-disease performance without restrictions) to 5 (dead). Change was day 28 minus baseline.
Time Frame: Baseline, Day 28 or ET
Population: Data not analyzed due to early study termination.
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Pregabalin | Placebo
Serious Adverse Events (participants affected / at risk) | 12/72 | 12/80
Other Adverse Events (participants affected / at risk) | 38/72 | 31/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=72) | Placebo (N=80)
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Device dislocation (General disorders) | 1 | 0
Disease progression (General disorders) | 4 | 3
Malaise (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 1
Septic shock (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Metabolic disorder (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=72) | Placebo (N=80)
Vertigo (Ear and labyrinth disorders) | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 3
Nausea (Gastrointestinal disorders) | 7 | 10
Vomiting (Gastrointestinal disorders) | 6 | 4
Fatigue (General disorders) | 8 | 4
Oedema peripheral (General disorders) | 4 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 2
Disturbance in attention (Nervous system disorders) | 4 | 0
Dizziness (Nervous system disorders) | 11 | 7
Headache (Nervous system disorders) | 4 | 2
Somnolence (Nervous system disorders) | 18 | 6
Tremor (Nervous system disorders) | 5 | 2
Dysuria (Renal and urinary disorders) | 0 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 2

LIMITATIONS AND CAVEATS:
Efficacy parameters baseline=the last non-missing observation, up to the baseline visit for that efficacy parameter. Baseline mBPI scores=average score in week preceding randomization, minimum 4 datapoints. No formal hypothesis testing conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.